CLINICAL TRIAL: NCT03839628
Title: Translational Control of Anabolic Resistance in Aging Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Micah Drummond, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Leucine study; R21AR073422 (NIH)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be tested before and 2-weeks after they have reduced their level of physical activity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced Physical Activity (Experimental): Participants will reduce their physical activity levels for 2-weeks by approximately 75% of their baseline level of physical activity
  Interventions: Other: Reduced Physical Activity

INTERVENTIONS:
Other: Reduced Physical Activity — Participants will reduce their level of physical activity for 2-weeks as defined as approximately 75% reduction from their baseline level of physical activity.
  Other Names: Muscle Disuse

SUMMARY:
This is an interventional study enrolling older individuals aged 60-85y to observe changes during physical inactivity. This study is investigating the relation between short-term physical inactivity and the impact of muscle health and function. The enrollment goal is 8 participants. The study will occur over the course of a month where participants will undergo testing before and after a reduction in physically activity levels. There will be a screening event collecting baseline data, two body composition scans, muscle function and oral glucose tolerance tests and a metabolic study before and after a 2-week period of inactivity. Each metabolic study will entail three-muscle biopsies: one before and 2 after the ingestion of leucine.

DETAILED DESCRIPTION:
Pre-testing- The baseline evaluation will assess muscle function and strength, and an oral glucose tolerance test. After the baseline visit, participants will be provided with a step activity monitor to track their level of activity. This will provide a baseline of the participant's normal level of physical activity so an accurate level of 75% activity reduction can be determined. A 3-day daily dietary diary will be provided for the participant to self-report prior to the experiment, as well.

Day 1- After the participant completes their normal activity log and dietary diary, they will be asked to return to the research center for a body composition scan and a metabolic study.

The metabolic study will involve blood sampling from an arm vein and muscle biopsies from the thigh before and after a leucine drink.

2-week period of inactivity- After the metabolic study, the participant will return home and maintain a reduced level of activity (75% reduction) for a two-week period. During this time, the participant will receive phone calls from research personnel in order to maintain adherence to the intervention.

Day 14- After the 2-week reduced activity period, the participant will return to the research center to receive a body composition scan and undergo a metabolic study identical to 'Day 1'.

Post-testing- After Day 14, the participant will be asked to return once again to the research center for a oral glucose tolerance test and the exercise lab for muscle function testing.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-85 years
* Ability to sign informed consent
* Free-living, prior to admission

Exclusion Criteria:

* Cardiac abnormalities considered exclusionary by the study physician (e.g., Chronic heart Failure, right-to-left shunt)
* Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
* History of kidney disease or failure
* Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
* Risk of blood clotting including family history of thrombophilia, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocystinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombine III
* Use of anticoagulant therapy (e.g., Coumadin, heparin)
* Elevated systolic pressure >150 or a diastolic blood pressure > 100
* Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
* Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
* Currently on a weight-loss diet or body mass index > 30 kg/m2
* Chronic systemic corticosteroid use (≥ 2 weeks) within 4 weeks of enrollment and for study duration (intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids are permitted). Androgens or growth hormone within 6 months of enrollment and for study duration (topical physiologic androgen replacement is permitted)
* History of stroke with motor disability
* A recent history (<12 months) of GI bleed
* History of liver disease
* History of respiratory disease (acute upper respiratory infection, history of chronic lung disease)
* Prior history of Heparin-Induced Thrombocytopenia
* An HbA1c value at or greater than 6.5%
* Any other condition or event considered exclusionary by the PI and faculty physician

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No plan has been put into place

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Physical Activity
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Physical Activity
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
HbA1c [Mean (Standard Deviation); unit: % of hemoglobin] | 5.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Lean Mass
Description: Change in lean mass
Time Frame: baseline and 2-weeks
Measure: Mean (Standard Error); unit: grams
Arm/Group | Reduced Physical Activity
Number analyzed (Participants) | 9
grams | 403 (142)

2. Primary Outcome: Strength
Description: Change in muscle strength
Time Frame: baseline and 2-weeks
Measure: Mean (Standard Error); unit: percentage of leg strength
Arm/Group | Reduced Physical Activity
Number analyzed (Participants) | 9
percentage of leg strength | -8 (.1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Reduced Physical Activity
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03839628/Prot_000.pdf